CLINICAL TRIAL: NCT02677467
Title: Epistaxis Correlate With Cardiovascular Disease?
Brief Title: Correlation Between Epistaxis and Cardiovascular Disease
Acronym: CBECD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, LEE YOON-JE, Fellowship, Emergency Medincine, Hanyang University
Other Study IDs: Gurivengers
Record Dates: First submitted 2016-01-31; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Disease; Epistaxis
MeSH Terms: conditions — Cardiovascular Diseases; Epistaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Blood sample for evaluating about cardiovasular risk.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Spontaneous epistaxis: A participant enroll if their age is over 18 with spontaneous epistaxis and their cause of visiting ER is spontaneous epistaxis. Exclusion criteria is that they needs immediately treatment for hypertensive urgency. And, they don't want to participate in this investigation. Investigators examine their blood-pressure variability and cardiovascular risk throughout their blood sample analysis.
  Interventions: Biological: Blood-pressure variability
- Bleeding of wound: A participant enroll if their age is over 18 with bleeding of wound and their cause of visiting ER is to bleed on wound. Exclusion criteria is that their wounds' condition is serious or their pain is much severe. And, they don't want to participate in this investigation. Investigators examine their blood-pressure variability and cardiovascular risk throughout their blood sample analysis.
  Interventions: Biological: Blood-pressure variability

INTERVENTIONS:
Biological: Blood-pressure variability — Day to Night Blood pressure variability

SUMMARY:
Investigators examine blood-pressure variance, several cardiovascular risk factors of patient with epistaxis. As a result of collected data, investigators look into correlation between epistaxis and hypertensive cardiovascular disorder.

DETAILED DESCRIPTION:
This study is prospective observational single blinded study.

A participant is visit in the ER who patient with epistaxis.

Investigators will enroll 50 patients with epistaxis. Exclusion criteria is that patient needs immediately treatment for hypertensive urgency or patient with nasal trauma.

Investigators examine blood-pressure (BP) at five times in Emergency Department (ED) and out-patient department (opd) of Otorhinolaryngology (OL) . Investigators explain this study and ask to write consent for participant. After proper management of epistaxis, investigators get blood sampling of the participant and, the participant has a reservation to "opd of cardiovascular division of Internal Medicine" (CV opd) in the hospital.

When the participant visit CV opd, the participant undergo 24-hours-BP-monitoring and Pulse wave velocity (PWV).

After that, the participant will be follow-up for 3 months.

Investigators collect 50 data from 50 participants as a registry and analyze the data.

ELIGIBILITY:
Group A

Inclusion Criteria:

* age is over 18 with spontaneous epistaxis

Exclusion Criteria:

* they needs immediately treatment for hypertensive urgency.
* they don't want to participate in this investigation.

Group B

Inclusion Criteria:

* age is over 18 with bleeding of wound

Exclusion Criteria:

* their wounds' condition is serious or their pain is much severe.
* they don't want to participate in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A : A participant enroll if their age is over 18 with spontaneous epistaxis and their cause of visiting ER is spontaneous epistaxis. Exclusion criteria is that they needs immediately treatment for hypertensive urgency. And, they don't want to participate in this investigation.
  Group B : A participant enroll if their age is over 18 with bleeding of wound and their cause of visiting ER is to bleed on wound. Exclusion criteria is that their wounds' condition is serious or their pain is much severe. And, they don't want to participate in this investigation.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Cholesterol level in each group | 1 day
BP variability level in each group | 1 day
Pulse wave velocity in each group | 1 day

SECONDARY OUTCOMES:
Smoking History in each group | 1 day
  Example = "12 pack-year"
Body Mass Index in each group | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: JUNGHOON SHIN, M.D., Ph.D., Study Chair — Hanyang University Guri Hospital
Locations (1):
- Hanyang University Guri Hospital, Guri-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The investigators make a registry for individual participant data and collect the registry and share it.